CLINICAL TRIAL: NCT07199556
Title: Study of the Impact of a Nutraceutical on Pain in Women With Musculoskeletal Symptoms Associated With Hormonal Therapy With Aromatase Inhibitors, in ER and/or PgR Positive Breast Cancer, After Antitumor Therapy.
Brief Title: Impact of a Food Supplement on Musculoskeletal Pain in Women With Breast Cancer Treated With Aromatase Inhibitors.
Acronym: DOLFLEX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Arafarma Group, S.A. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ARA-EXP/TEN-2023-01
Record Dates: First submitted 2025-09-22; First posted 2025-09-30 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Dietary Supplements

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental): There is only one arm in the study. All patients will be treated with the experimental food supplement.
  Interventions: Dietary Supplement: Food supplement

INTERVENTIONS:
Dietary Supplement: Food supplement — Tenflex® is an authorized food supplement.

SUMMARY:
The aim of this pilot study is to assess the change in pain, measured with the Modified Brief Pain Inventory - Short Form (mBPI-sf), at 4, 8, and 12 weeks. The collagen- and chondroitin sulfate-based food supplement may help improve pain in these patients with musculoskeletal symptoms associated with hormone therapy in ER- and/or PR-positive breast cancer.

DETAILED DESCRIPTION:
ER- and/or PR-positive breast cancer is treated with hormone therapy. There is a relationship between the administration of hormone therapy and the presence and/or exacerbation of joint pain in patients with breast cancer.

The administration of food supplement may result in an improvement of pain, as measured by the mBPI-sf questionnaire, in patients undergoing treatment with Aromatase Inhibitors.

ELIGIBILITY:
Inclusion Criteria:

* Women with histologically confirmed hormone receptor-positive breast carcinoma, without evidence of metastatic disease (M0).
* Surgical treatment completed and any surgery-related complications resolved.
* Currently receiving hormonal therapy with aromatase inhibitors (AIs) for at least 21 days, with pain symptoms lasting less than 6 months attributable to AIs, and with a treatment plan to continue for at least an additional 180 days (6 months).
* Musculoskeletal symptoms associated with hormonal therapy that began or worsened after initiation of such therapy. New musculoskeletal pain must not be specifically due to fractures or traumatic injuries.
* "Average pain" score of at least 4, as assessed by the mBPI-sf questionnaire within 7 days prior to enrollment or baseline visit.
* ECOG performance status of 0-2.
* Patients able to provide informed consent.

Exclusion Criteria:

* Concurrent medical or arthritic conditions that may confound or interfere with the assessment of pain or efficacy, such as rheumatologic/inflammatory arthritis (rheumatoid arthritis, systemic lupus, spondyloarthropathy, psoriatic arthritis, polymyalgia rheumatica) or cancer that may affect bone.
* Chemotherapy and/or radiotherapy completed within 28 days prior to enrollment or baseline visit, and/or unresolved Grade ≥2 side effects related to chemotherapy and/or radiotherapy, except for alopecia and peripheral neuropathy.
* Known allergy or hypersensitivity to Tenflex®.
* Pregnant or breastfeeding patients.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2024-03-14 (Actual); Primary Completion 2025-07-21 (Actual); Study Completion 2025-09-10 (Actual)

PRIMARY OUTCOMES:
Change in average pain intensity modified Brief Pain Inventory - Short Form (mBPI-sf). | Baseline visit, Week 4 visit, Week 8 visit, Week 12 visit and Week 24 visit.
  To evaluate the change in average pain intensity as measured by the modified Brief Pain Inventory-Short Form (mBPI-sf) from baseline to Weeks 4, 8, 12, and 24 of treatment with Tenflex. It contains 11 items and these score 0 to 10 being higher the worse pain.

SECONDARY OUTCOMES:
Change in quality of life Short Form 12-Item Health Survey (SF-12). | Baseline visit, Week 4 visit, Week 8 visit, Week 12 visit and Week 24 visit.
  To evaluate the change of the quality of life questionnaire SF-12 from baseline to Weeks 4, 8, 12, and 24 of treatment with Tenflex. This survey measures eight health domains (Physical Functioning (PF), Role Physical (RP), Bodily Pain (BP), General Health (GH), Vitality (VT), Social Functioning (SF), Role Emotional (RE), Mental Health (MH)), which are summarized into two components summary scores: Physical Component Summary (PCS) and Mental Component Summary (MCS). Higher scores are better health status.
Change in quality of life 'BREAST-Q Reconstruction/Reduction/Augmentation Module'. | Baseline visit, Week 4 visit, Week 8 visit, Week 12 visit and Week 24 visit.
  To evaluate the change of the quality of life questionnaire Breast-Q from baseline to Weeks 4, 8, 12, and 24 of treatment with Tenflex. It contains differents scales and their raw scores are converted into a scale from 0 (worst possible outcome) to 100 (best possible outcome).
Percentage of patients with ≥30% reduction in average pain. | Baseline visit, Week 4 visit, Week 8 visit, Week 12 visit and Week 24 visit.
  To calculate the percentage of patients with 30% reduction in average pain from baseline to Weeks 4, 8, 12, and 24 of treatment with Tenflex.
Changes in other mBPI-sf domains. | Baseline visit, Week 4 visit, Week 8 visit, Week 12 visit and Week 24 visit.
  To evaluate changes in other mBPI-sf domains (general activity, mood, walking ability, normal work, relations with others, sleep, enjoyment of life) from baseline to Weeks 4, 8, 12, and 24.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Clínic Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided